CLINICAL TRIAL: NCT03843697
Title: A Controlled Trial for the Prevention of Loss of the Effect of Biological Drugs in Patients With Inflammatory Bowel Disease
Brief Title: A Trial for Prevention of Loss of the Effect of Biological Drugs in Patients With Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tahel Ilan Ber (Industry)
Responsible Party: Sponsor-Investigator, Tahel Ilan Ber, Chief Medical Officer, Oberon Sciences LTD
Organization: Oberon Sciences LTD (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: OS-002
Record Dates: First submitted 2018-12-21; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: The study will assess the effect of adding an app which reminds to take an approved therapy in patients who are already on the drug without a change of the physician's predetermined regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with IBD who develop resistance to anti TNF (Experimental): Patients with inflammatory bowel disease who developed partial or complete resistance to anti TNF based drugs
  Interventions: Device: An App for reminding patients to take their medication

INTERVENTIONS:
Device: An App for reminding patients to take their medication — Open-label, single-center study, up to 20 adults (>18) male and female with inflammatory bowel disease (chorn's disease, ulcerative colitis), unresponsive to biological drugs, will participate in a 4-week observation period during which no change in drugs is permitted. The patients will then begin 10-week treatment by taking their medications according to a semi-random schedule that is pre-set for them by the physician using the same drugs the patient is taking and only changing the dose and times of taking them each day while keeping the drugs within their therapeutic window.
  Other Names: Oberon APP

SUMMARY:
Trial for IBD patients non-responsive to biological drugs, using medical app reminding patients to take their physician-prescribed medications

DETAILED DESCRIPTION:
Patients with IBD who developed loss of response to anti-TNF based medications will receive a cell phone based app that will remind them to take the drug with an approved dosing range.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD or UC according to validated criteria, with a Crohn's Disease Activity Score (CDAI) of 200-450 at inclusion.
2. Patients on a stable dose within the last 6 weeks of any type of anti TNF agent or any other biological agent
3. 5-ASA (mesalamine), and immunomodulatory, or immunosuppressive agent, and symptomatic relief (anti-diarrheals) for patients are allowed in a stable dose (6 weeks).
4. Non-smoking (by declaration) for a period of at least 6 months.
5. Females of childbearing potential must be non-pregnant (as determined by a serum pregnancy test at screening and again, prior to each dosing session) and agree to use adequate contraceptive means throughout the study.
6. No known history of significant neurological, renal, cardiovascular, respiratory (asthma), endocrinological, gastrointestinal, primary hematopoietic disease, neoplasm, or any other clinically significant medical disorder other than Crohn's disease and its complications, which in the investigator's judgment contraindicate administration of the study medications.
7. No history of drug or alcohol abuse.
8. Screening tests must meet the following criteria: HGB ≥8.5 g/dL, platelets ≥ 100,000/ mm³, WBC: 3500-12,000/mm³, serum albumin above 2.5 g/dL, amylase, lipase and total bilirubin within normal limits. ALT, AST, alkaline phosphatase up to 1.5 times normal limits.
9. No clinically significant abnormalities in screening physical exam.
10. Negative HIV, Hepatitis B and Hepatitis C serology tests within 2 years.
11. Patients must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
12. Patients must satisfy a medical examiner about their fitness to participate in the study.
13. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients with evidence of other serious infectious, autoimmune, hepatic, nephritic or systemic disease or compromised organ function.
2. Patients with a present colostomy, ileostomy or subtotal colectomy with ileorectal anastomosis.
3. Symptomatic stenosis or ileal strictures, x-ray evidence of fibrosed bowel.
4. Patients presenting with, or with a history of persistent intestinal obstruction, bowel perforation, uncontrolled GI bleed or abdominal abscess or infection, toxic megacolon.
5. Patients with fistulating CD.
6. Short bowel syndrome.
7. Patients with a history of GI tract malignancy or IBD-associated malignant changes in the intestines.
8. Patients with any clinically significant abnormality upon physical examination or in the clinical laboratory test values.
9. A change in the dose of the immunomodulatory or immunosuppressive drug within 6 weeks.
10. Over-the-counter drugs, including herbal medications, and prescription drugs (other than those listed above) are not allowed for 7 days prior to first study dosing and throughout the duration of the study
11. Receipt of packed RBC's within 3 months prior to the first study dosing and throughout the study.
12. Participation in another clinical trial within 30 days prior to first drug administration.
13. Patients with an inability to communicate well with the PI and staff (i.e., language problem, poor mental development or impaired cerebral function).
14. Patients with any acute medical situation (e.g. acute infection) within 48 hours of first dosing session, which is considered of significance by the Principal Investigator.
15. Patients who will be unavailable for the duration of the trial, are likely to be noncompliant with the protocol, or who are felt to be unsuitable by the PI for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with reduction chron's disease activity index score more than 100 points during the study; | 10 weeks
  Proportion of subjects with reduction chron's disease activity index score more than 100 points during the study;

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical remission or response without steroid rescue therapy during the study; | 10 weeks
  The secondary efficacy outcome was the proportion of subjects with clinical response at week 10

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azmanov H, Ross EL, Ilan Y. Establishment of an Individualized Chronotherapy, Autonomic Nervous System, and Variability-Based Dynamic Platform for Overcoming the Loss of Response to Analgesics. Pain Physician. 2021 May;24(3):243-252. PMID 33988944